CLINICAL TRIAL: NCT02373969
Title: Thromboelastogram During Surgery for Total Knee Replacement With Tourniquet Application and Single Dose Tranexamic Acid
Brief Title: Thromboelastogram During Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: TEG-099-11
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Orthopedic Procedures, Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Verify the changes in coagulation system during total knee replacement surgery with tranexamic acid single bolus infusion.

DETAILED DESCRIPTION:
The study was set to reveal changes in the coagulation and fibrinolytic systems during total knee surgery and especially during tourniquet placement, tourniquet removal and revascularization of ischemic limb, after tranexamic acid single bolus infusion, and at post operative day 1.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* TKR operation elective
* ASA I-III

Exclusion Criteria:

* TKR due to any reason but osteoarthrosis
* known coagulation problems
* platelets < 100,000/DcL
* Hb < 12 g%
* past thrombo-embolic event
* treatment with aspiring during last week
* treatment with NSAID's during last 48 hours
* malignancy
* known allergy to tranexamic acid
* general anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As described in eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in coagulation status during and after surgery compared to pre-surgery | During and after surgery compared to pre-surgery
Change in fibrinolytic activity during and after surgery compared to pre-surgery | During and after surgery compared to pre-surgery

IPD SHARING:
Plan to Share IPD: No